CLINICAL TRIAL: NCT00560820
Title: Phase I Study to Examine the Effect of Deferasirox on Renal Hemodynamics in β-thalassemia Patients With Transfusional Iron Overload
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2123; 2006-006838-17 (EudraCT Number)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2016-06

CONDITIONS: β-thalassemia; Transfusional Iron Overload
Keywords: β-thalassemia; transfusional iron overload; renal function; renal biomarkers; deferasirox
MeSH Terms: interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox (Experimental): 30 mg/kg/day
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — 30 mg/kg/day
  Other Names: ICL670

SUMMARY:
The primary purpose of this study is to evaluate the effect of deferasirox on renal hemodynamics by determining glomerular filtration rate (GFR), renal plasma flow (RPF) and filtration fraction (FF).

ELIGIBILITY:
Inclusion criteria:

* Male or female patients ≥ 18 years of age without prior history of deferasirox treatment
* β-thalassemia patients receiving regular transfusions every 2-5 weeks
* Transfusion history of ≥ 20 units of packed red blood cells

Exclusion criteria:

* Abnormal renal function at baseline
* ALT greater than 5 x ULN at screening
* Patients with underlying cardiac disease requiring continuous iron chelation therapy

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Effect of deferasirox on renal hemodynamics in patients with β-thalassemia and transfusional iron overload. | Once a month

SECONDARY OUTCOMES:
Effect of deferasirox on standard markers of renal function | Once a month

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (3):
- Italy (3):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Orbassano

REFERENCES:
- [Derived] Piga A, Fracchia S, Lai ME, Cappellini MD, Hirschberg R, Habr D, Wegener A, Bouillaud E, Forni GL. Deferasirox effect on renal haemodynamic parameters in patients with transfusion-dependent beta thalassaemia. Br J Haematol. 2015 Mar;168(6):882-90. doi: 10.1111/bjh.13217. Epub 2014 Nov 17. PMID 25402221
- See also: Results for CICL670A2123 can be found on the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7823